CLINICAL TRIAL: NCT01976884
Title: Expression and the Clinical Significance of Neutrophil PD-L1 During Sepsis
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Jia-feng Wang, Dr., Changhai Hospital
Other Study IDs: NeutrophilPD-L1
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-10

CONDITIONS: Sepsis; Immunosuppression
Keywords: sepsis; immunosuppression; PD-L1
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood sample was collected for detection of neutrophil PD-L1, monocyte HLA-DR and lymphocyte PD-1.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Severe sepsis: Patients with severe sepsis
- Infectious kidney stone: Patients with sepsis after PCNL for infectious kidney stone
- Tumor: Patients with pancreatic cancer
- Volunteer

SUMMARY:
Immunosuppression is the leading cause of death in septic patients. Neutrophils are classical components of innate immunology, but recent studies showed that neutrophils might display antigen presenting function and inhibit lymphocyte proliferation by expressing programmed cell death 1 ligand 1 (PD-L1). Whether neutrophils express PD-L1 and its role in immunosuppression during sepsis remain unclear.

ELIGIBILITY:
Inclusion Criteria:

* patients with severe sepsis
* patients with sepsis after PCNL for infectious kidney stone
* patients with pancreatic cancer
* healthy volunteers

Exclusion Criteria:

* patients with immunodeficient diseases
* patients who accept glucocorticoid or immunosuppressant
* patients with an age older than 18 years
* patients providing the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted in ICU at Changhai Hospital
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
PD-L1 level on neutrophils | within 24h after recruitment
  PD-L1 level on neutrophils was compared between different populations.

SECONDARY OUTCOMES:
28-day mortality | 28 days after diagnosis of sepsis